CLINICAL TRIAL: NCT00655746
Title: The Effect of Omeprazole on the Pharmacokinetics of Dasatinib (BMS-354825) in Healthy Subjects
Brief Title: The Effect of Omeprazole on the Pharmacokinetics of Dasatinib in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CA180-249
Record Dates: First submitted 2008-04-03; First posted 2008-04-10 (Estimated); Results first posted 2009-07-31 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Healthy
Keywords: Healthy Subjects
MeSH Terms: interventions — Dasatinib; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Dasatinib + Omeprazole

INTERVENTIONS:
Drug: Dasatinib + Omeprazole — Tablet/Capsule, Oral, (Dasatinib 100 mg)/(Omeprazole 40 mg), once daily, 7 days
  Other Names: Sprycel

SUMMARY:
The purpose of this study is to assess the effect of omeprazole on the pharmacokinetics of dasatinib in healthy subjects and to assess the safety and tolerability of a single dose of dasatinib before and after 5 days of dosing with omeprazole in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by medical history, physical examination, ECGs, and clinical laboratory determinations

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Prior exposure to dasatinib

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2008-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bristol-Myers Squibb Clinical Pharmacology Unit, Hamilton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 49 participants were enrolled in the study, and 35 discontinued before being treated (26 no longer met study criteria, 6 withdrew consent, 3 group full/not needed)
Groups:
- Dasatinib/Omeprazole: Day 1: 100-mg oral dasatinib; Days 2 through 6: 40-mg oral omeprazole; Day 6:100-mg oral dasatinib and 40-mg oral omeprazole
Period: Overall Study
Arm/Group | Dasatinib/Omeprazole
Started | 14
Completed | 13
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib/Omeprazole
Number analyzed (Participants) | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 37 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 8
  White | 5
  Asian | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 25.4 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Dasatinib Pharmacokinetic (PK) Parameter: Maximum Observed Plasma Concentration (Cmax)
Description: Pharmacokinetics is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. Cmax=maximum observed plasma concentration of dasatinib
Time Frame: Day 1 and Day 6 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours post dose
Measure: Geometric Mean (Full Range); unit: ng/mL
Groups:
- Dasatinib (Day 1): 100-mg oral dasatinib
- Dasatinib + Omeprazole (Day 6): 100-mg oral dasatinib and 40-mg oral omeprazole
Arm/Group | Dasatinib (Day 1) | Dasatinib + Omeprazole (Day 6)
Number analyzed (Participants) | 14 | 13
ng/mL | 65.58 (51) [3.17 to 150.81] | 38.64 (76) [1.96 to 146.78]

2. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths and Discontinuations
Description: An AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a patient or clinical investigation subject administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: At Informed Consent (within 21 days of Day 1) through Study Discharge (Day 7)
Measure: Number; unit: Participants
Groups:
- Omeprazole (Days 2-5): 40-mg oral omeprazole
Arm/Group | Dasatinib (Day 1) | Omeprazole (Days 2-5) | Dasatinib + Omeprazole (Day 6) | All Participants
Number analyzed (Participants) | 14 | 14 | 13 | 14
Participants
  Number of Participants with ≥1 AE | 3 | 2 | 2 | 4
  Death | 0 | 0 | 0 | 0
  SAE | 0 | 0 | 0 | 0
  Discontinuation due to AEs | 0 | 0 | 0 | 0

3. Primary Outcome: Dasatinib PK Parameter Time of Maximum Observed Plasma Concentration(Tmax)
Description: Pharmacokinetics is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. Tmax=time of maximum observed plasma concentration
Time Frame: Day 1 and Day 6 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours post dose
Measure: Median (Full Range); unit: hours
Arm/Group | Dasatinib (Day 1) | Dasatinib + Omeprazole (Day 6)
Number analyzed (Participants) | 14 | 13
hours | 0.75 [0.47 to 2.02] | 1.00 [0.50 to 1.92]

4. Primary Outcome: Dasatinib PK Parameter: Plasma Half-Life (T-HALF)
Description: Pharmacokinetics is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. T-Half=plasma half-life
Time Frame: Day 1 and Day 6 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours post dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dasatinib (Day 1) | Dasatinib + Omeprazole (Day 6)
Number analyzed (Participants) | 14 | 13
hours | 4.00 (1.35) | 4.29 (1.62)

5. Primary Outcome: Dasatinib PK Parameter: Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC[0-T])
Description: area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC[0-T])for dasatinib
Time Frame: Day 1 and Day 6 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours post dose
Measure: Geometric Mean (Full Range); unit: ng∙h/mL
Arm/Group | Dasatinib (Day 1) | Dasatinib + Omeprazole (Day 6)
Number analyzed (Participants) | 14 | 13
ng∙h/mL | 249.46 [42.42 to 531.26] | 137.49 [14.03 to 453.41]

6. Primary Outcome: Dasatinib PK Parameters: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinite Time (AUC[INF])
Description: Pharmacokinetics is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. AUC(INF)=area under the plasma concentration-time curve from time zero extrapolated to infinite time
Time Frame: Day 1 and Day 6 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 24 hours post dose
Measure: Geometric Mean (Full Range); unit: ng∙h/mL
Arm/Group | Dasatinib (Day 1) | Dasatinib + Omeprazole (Day 6)
Number analyzed (Participants) | 14 | 13
ng∙h/mL | 265.40 [51.18 to 542.97] | 152.84 [19.61 to 460.78]

ADVERSE EVENTS:
Arm/Group | BMS-354825 + Omeprazole
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 4/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-354825 + Omeprazole (N=14)
HEADACHE (Nervous system disorders) | 3
NAUSEA (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
FLATULENCE (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.